CLINICAL TRIAL: NCT02021305
Title: The Role of TLR-4 Asp299Gly and Thr399Ile Polymorphisms in Children With Urinary Tack Infections
Brief Title: The Role of TLR-4 Polymorphisms in Children With Urinary Track Infections
Acronym: TLR-4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Panagiota Karananou, MD, Aristotle University Of Thessaloniki
Other Study IDs: 230283
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Urinary Tract Infection
Keywords: Toll like Receptors; TLR 4; Urinary track infections in children; TLR 4 polymorphisms; Innate immunity; Defence mechanisms; Immune responses
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: 60 children with a recorded episode of acute Urinary Track infection who attended 4th Department of Pediatrics of Medical School of Aristotle University of Thessaloniki.
- Controls: 100 children with no history of Urinary Track Infection who attended 4th Department of Pediatrics of Medical School of Aristotle University of Thessaloniki.

SUMMARY:
Purpose So far anatomical abnormalities (mostly congenital) were, in the majority of the patients, associated with urinary track infections. In this study the researchers will try to investigate the role of TLRs as molecular interactions between bacterial virulence and host response.

TLRs are important mediators in the development of the natural immunity against bacteria. They recognize microbial pathogen associated molecular patterns and alert the host's immune system to the presence of invading microbes

DETAILED DESCRIPTION:
The aim of his observational case-control study is to :

1. investigate if the expression of TLR2 and TLR4 mediate in the development of the natural immunity of the uroepithileal cells against bacteria.
2. evaluate the effect of the TLR-gene Asp299Gly and Thr399Ile polymorphisms on the development and clinical severity of urinary tract infections (UTI) in children.
3. determine the association of the expression of TLR-2 and TLR-4 and TLR-4 polymorphisms with the formation of renal scar in children.
4. investigate the expression of TLR-2 and TLR-4 and TLR-4 polymorphisms in healthy children and elaborate the results to the possible carriers of these polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* For the patients

  * 6months -14 years of age
  * unrelated male and female children with one episode of acute urinary track infection (positive urine culture and clinical symptoms )
  * with/without anatomic genitourinary anomalies .
  * children with upper UTI or children with lower UTI
  * Sign written informed consent

Inclusion Criteria:

For the controls

* 6 months-14 years of age
* age and gender matched with the patients
* unrelated male and female children with no recorded history of urinary track infection and negative urine cultures .
* Sign written informed consent

Exclusion Criteria:

* For the patients

  * Subjects who do not meet the criteria above
  * Severe or chronic illness
  * Symptoms of acute infection
  * Immune deficiency or immune suppressor therapy
  * Medication

Exclusion Criteria:

For the controls

* Subjects who do not meet the criteria above
* Severe or chronic illness
* Symptoms of acute infection
* Immune deficiency or immune suppressor therapy
* Medication

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients an controls are selected from the Emergency Department and Outpatient Clinics of the 4th Department of Pediatrics , Aristotle University of Thessaloniki, Papageorgiou Hospital, Thessaloniki, Greece
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
frequency of TLR-4 299, 399 polymorphism and expression of TLR-2 and TLR-4 by monocytes in children with urinary track infection and healthy controls. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Efimia Papadopoulou-Alataki, MD, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Thessaloniki, Greece